CLINICAL TRIAL: NCT00716079
Title: An International Randomised Controlled Trial to Establish the Effects of Early Intensive Blood Pressure Lowering in Patients With Intracerebral Haemorrhage.
Brief Title: The Second Intensive Blood Pressure Reduction in Acute Cerebral Haemorrhage Trial
Acronym: INTERACT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Craig Anderson, Senior Director, Neurological and Mental Health Division, The George Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHMRC-571281
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Intracerebral Hemorrhage; Stroke; Hypertension
Keywords: Cerebral Hemorrhage; Stroke; antihypertensive drugs; blood pressure; disability; clinical trial; outcomes
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hypertension | interventions — Labetalol; Metoprolol; Hydralazine; Nitroglycerin; Phentolamine; Nicardipine; urapidil; esmolol; Clonidine; Enalaprilat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive BP lowering (Other): Management policy to lower the systolic Blood pressure (BP) to a target of 140mmHg within 1 hour of randomization and sustained for 24 hours. Sites were provided with protocols for different intravenous agents and used whichever routinely available drugs were in their hospital.
  Interventions: Other: Blood pressure management policies
- Guideline recommended BP lowering (Other): Patients received management of BP based on the standard guidelines at the time, as published by the American Heart Association (AHA) in 2007 and 2010. The attending clinician may consider commencing BP treatment if the systolic level is greater than 180 mmHg, however and the first line treatment will be oral (including nasogastric if required) and/or transdermal routes. Should control of systolic BP not be achieved via these routes, intravenous treatment may be started until the target systolic BP of 180 mmHg is achieved.
  Interventions: Other: Blood pressure management policies

INTERVENTIONS:
Other: Blood pressure management policies — The trial is an assessment of BP lowering management strategies, using routinely available drugs. There is some flexibility in the use of particular BP lowering agents to achieve BP targets.
  Other Names: Labetalol Hydrochloride; Metoprolol tartrate; Hydralazine Hydrochloride; Glycerol Trinitrate; Phentolamine mesylate; Nicardipine; Urapidil; Esmolol; Clonidine; Enalaprilat; Niroprusside

SUMMARY:
The purpose of this academic lead study is to determine if a treatment strategy of early intensive blood pressure (BP) lowering compared to conservative BP lowering policy in patients with elevated blood pressure within 6 hours of acute intracerebral haemorrhage (ICH) improves the outcome of death and disability at 3 months after onset.

DETAILED DESCRIPTION:
Intracerebral haemorrhage (ICH) is one of the most serious subtypes of stroke, affecting over a million people worldwide each year, most of whom live in Asia. About one third of people with ICH die early after onset and the majority of survivors are left with major long-term disability. Despite the magnitude of the disease burden and cost on healthcare resources, there remains uncertainty about the role of surgery for ICH and no acute medical therapies have been shown to definitely alter outcome in ICH.

The INTERACT2 study follows the recently completed initial pilot study vanguard phase) which established the feasibility of the protocol, safety of early intensive BP lowering, and effects on haematoma expansion within 6 hours of onset of ICH. Having established 'proof-of-concept' that BP lowering may improve outcome by reducing haematoma expansion, INTERACT2 aims to establish the effects of the treatment on major clinical endpoints in patients with ICH recruited from an expanding clinical network around the world.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CT-confirmed spontaneous Intracerebral Haemorrhage (ICH)
* Elevated systolic blood pressure (>150mmHg and <220mmHg)
* Capacity to commence randomly assigned treatment within 6 hours of onset of ICH.
* Able to be 'actively' treated and admitted to a monitored facility

Exclusion Criteria:

* Clear indication or contraindication to intensive BP lowering.
* Evidence ICH secondary to a structural abnormality
* Use of thrombolytic agent
* Previous ischaemic stroke within 30 days
* A very high likelihood that the patient will die within the next 24 hours on the basis of clinical and/or radiological criteria
* Score of 3-5 on the Glasgow Coma Scale (indicating deep coma)
* Significant pre-stroke disability or advanced dementia
* Planned early neurological intervention
* Participation in another clinical trial.
* A high likelihood that the patient will not adhere to the study treatment and follow-up regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2839 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, PhD, Principal Investigator — The George Institute
Locations (62):
- Mayo Clinic, Rochester, Minnesota, United States
- Regional Coordinating Centre Argentina, Buenos Aires, Argentina
- Australia (12):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Concord Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital Health Service District, Brisbane, Queensland
  - Western Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Austin Repatriation General Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Austria (3):
  - University of Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - Allgemeines Krankenhaus Linz, Linz
- Belgium (2):
  - AZ-VUB (University hospital Brussels), Jette
  - CHU Tivoli, La Louvière
- Regional Coordinating Centre Brazil, São Paulo, Brazil
- Regional Coordnating Centre Chile, Santiago, Chile
- China (2):
  - Regional Coordinating Centre China: The George Institute China, Beijing, Beijing Municipality
  - Regional Coordinating and Monitoring Centre: Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai Institute of Hypertension, Shanghai Second Medical University, Shanghai
- Helsinki University Central Hospital, Helsinki, Finland
- France (15):
  - Hôpital Jean Minjoz, Besançon
  - Hopital de la Cavale-Blanche, Brest
  - Centre Hospitalier de Calais, Calais
  - CHU Bicetre, Le Kremlin-Bicêtre
  - Hopital Roger Salengro, Lille
  - Centre Hospitalier de Meaux, Meaux
  - CHU Nantes - Hopital Laennec, Nantes
  - Hopital de Lariboisiere, Paris
  - Centre Hospitalier Sainte Anne, Paris
  - Regional Coordinating Centre Europe: Unite de recherche clinique Lariboisiere, Paris
  - Hôpital de la Salpêtrière, Paris
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Hopital Tenon, Paris
  - Hopital Delafontaine, Saint-Denis
  - Centre Hospitalier de Versailles, Versailles
- Germany (13):
  - Charite Campus Benjamin Franklin (CCBF), Berlin
  - Universitatsklinikum Dresden, Dresden
  - Heinrich-Heine-Universitat, Düsseldorf
  - Universitat Erlangen-Nurnberg, Erlangen
  - Klinikum Frankfurt, Frankfurt
  - Universitatsklinikum Frankfurt, Frankfurt
  - Martin-Luther-Universität, Halle
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - University of Heidelberg, Heidelberg
  - Universitatsklinikum Mannheim, Mannheim
  - Universitatsklinikum Ulm, Oberer Eselsberg, Ulm
- Prince of Wales Hospital, Shatin, Hong Kong
- Regional Coordinating Centre India: The George Institute India, Hyderabad, Andhra Pradesh, India
- Ospedale di Citta di Castello, Città di Castello, Italy
- The Aga Khan University Hospital, Karachi, Pakistan
- Hospital de Sao Joao, Porto, Portugal
- Spain (3):
  - Hospital General Universitario de Albacete, Albacete
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de Girona Dr. Josep Trueta, Girona
- Inselspital Neurologische Klinik, Bern, Switzerland
- Regional Coordinating Centre United Kingdom, Leicester, United Kingdom

REFERENCES:
- [Background] Anderson CS, Huang Y, Wang JG, Arima H, Neal B, Peng B, Heeley E, Skulina C, Parsons MW, Kim JS, Tao QL, Li YC, Jiang JD, Tai LW, Zhang JL, Xu E, Cheng Y, Heritier S, Morgenstern LB, Chalmers J; INTERACT Investigators. Intensive blood pressure reduction in acute cerebral haemorrhage trial (INTERACT): a randomised pilot trial. Lancet Neurol. 2008 May;7(5):391-9. doi: 10.1016/S1474-4422(08)70069-3. Epub 2008 Apr 7. PMID 18396107
- [Background] Delcourt C, Huang Y, Wang J, Heeley E, Lindley R, Stapf C, Tzourio C, Arima H, Parsons M, Sun J, Neal B, Chalmers J, Anderson C; INTERACT2 Investigators. The second (main) phase of an open, randomised, multicentre study to investigate the effectiveness of an intensive blood pressure reduction in acute cerebral haemorrhage trial (INTERACT2). Int J Stroke. 2010 Apr;5(2):110-6. doi: 10.1111/j.1747-4949.2010.00415.x. PMID 20446945
- [Derived] Wang X, Ren X, Li Q, Ouyang M, Chen C, Delcourt C, Chen X, Wang J, Robinson T, Arima H, Ma L, Hu X, You C, Li G, Jie Y, Lin Y, Billot L, Munoz-Venturelli P, Martins S, Pontes-Neto OM, Liu L, Chalmers J, Carcel C, Song L, Anderson CS; INTERACT Investigators. Effects of blood pressure lowering in relation to time in acute intracerebral haemorrhage: a pooled analysis of the four INTERACT trials. Lancet Neurol. 2025 Jul;24(7):571-579. doi: 10.1016/S1474-4422(25)00160-7. PMID 40541207
- [Derived] You S, Zheng D, Chen X, Wang X, Ouyang M, Han Q, Cao Y, Delcourt C, Song L, Carcel C, Arima H, Liu CF, Lindley RI, Robinson T, Anderson CS, Chalmers J; INTERACT Investigators. Subacute Neurological Improvement Predicts Favorable Functional Recovery After Intracerebral Hemorrhage: INTERACT2 Study. Stroke. 2025 Mar;56(3):621-627. doi: 10.1161/STROKEAHA.124.048847. Epub 2025 Feb 3. PMID 39895502
- [Derived] You S, Zheng D, Yoshimura S, Ouyang M, Han Q, Wang X, Cao Y, Delcourt C, Song L, Arima H, Chen X, Liu CF, Lindley RI, Robinson T, Anderson CS, Chalmers J; INTERACT Investigators. Optimum Baseline Clinical Severity Scale Cut Points for Prognosticating Intracerebral Hemorrhage: INTERACT Studies. Stroke. 2024 Jan;55(1):139-145. doi: 10.1161/STROKEAHA.123.044538. Epub 2023 Nov 29. PMID 38018833
- [Derived] Malavera A, You S, Zheng D, Delcourt C, Anderson CS; INTERACT2 Investigators. Prognostic significance of early pyrexia in acute intracerebral haemorrhage: The INTERACT2 study. J Neurol Sci. 2021 Apr 15;423:117364. doi: 10.1016/j.jns.2021.117364. Epub 2021 Feb 26. PMID 33647734
- [Derived] Sandset EC, Wang X, Carcel C, Sato S, Delcourt C, Arima H, Stapf C, Robinson T, Lavados P, Chalmers J, Woodward M, Anderson CS. Sex differences in treatment, radiological features and outcome after intracerebral haemorrhage: Pooled analysis of Intensive Blood Pressure Reduction in Acute Cerebral Haemorrhage trials 1 and 2. Eur Stroke J. 2020 Dec;5(4):345-350. doi: 10.1177/2396987320957513. Epub 2020 Sep 20. PMID 33598552
- [Derived] Song L, Wang X, Ouyang M, Sun L, Chen X, Arima H, Sandset EC, Delcourt C, Wang J, Chen G, Robinson T, Lindley RI, Chalmers J, Anderson CS; INTERACT2 Investigators. Associations of an Abnormal Physiological Score With Outcomes in Acute Intracerebral Hemorrhage: INTERACT2 Study. Stroke. 2021 Jan;52(2):722-725. doi: 10.1161/STROKEAHA.120.030435. Epub 2021 Jan 11. PMID 33423518
- [Derived] Wang X, Moullaali TJ, Li Q, Berge E, Robinson TG, Lindley R, Zheng D, Delcourt C, Arima H, Song L, Chen X, Yang J, Chalmers J, Anderson CS, Sandset EC. Utility-Weighted Modified Rankin Scale Scores for the Assessment of Stroke Outcome: Pooled Analysis of 20 000+ Patients. Stroke. 2020 Aug;51(8):2411-2417. doi: 10.1161/STROKEAHA.119.028523. Epub 2020 Jul 9. PMID 32640944
- [Derived] You S, Zheng D, Delcourt C, Sato S, Cao Y, Zhang S, Yang J, Wang X, Lindley RI, Robinson T, Anderson CS, Chalmers J. Determinants of Early Versus Delayed Neurological Deterioration in Intracerebral Hemorrhage. Stroke. 2019 Jun;50(6):1409-1414. doi: 10.1161/STROKEAHA.118.024403. Epub 2019 Apr 18. PMID 31136288
- [Derived] Wang X, Sandset EC, Moullaali TJ, Chen G, Song L, Carcel C, Delcourt C, Woodward M, Robinson T, Chalmers J, Arima H, Anderson CS; INTERACT2 Investigators. Determinants of the high admission blood pressure in mild-to-moderate acute intracerebral hemorrhage. J Hypertens. 2019 Jul;37(7):1463-1466. doi: 10.1097/HJH.0000000000002056. PMID 31085948
- [Derived] Chen R, Wang X, Anderson CS, Robinson T, Lavados PM, Lindley RI, Chalmers J, Delcourt C. Infratentorial Intracerebral Hemorrhage. Stroke. 2019 May;50(5):1257-1259. doi: 10.1161/STROKEAHA.118.023766. PMID 30890109
- [Derived] Moullaali TJ, Wang X, Martin RH, Shipes VB, Qureshi AI, Anderson CS, Palesch YY. Statistical analysis plan for pooled individual patient data from two landmark randomized trials (INTERACT2 and ATACH-II) of intensive blood pressure lowering treatment in acute intracerebral hemorrhage. Int J Stroke. 2019 Apr;14(3):321-328. doi: 10.1177/1747493018813695. Epub 2018 Nov 12. PMID 30418098
- [Derived] Delcourt C, Sato S, Zhang S, Sandset EC, Zheng D, Chen X, Hackett ML, Arima H, Hata J, Heeley E, Al-Shahi Salman R, Robinson T, Davies L, Lavados PM, Lindley RI, Stapf C, Chalmers J, Anderson CS; INTERACT2 Investigators. Intracerebral hemorrhage location and outcome among INTERACT2 participants. Neurology. 2017 Apr 11;88(15):1408-1414. doi: 10.1212/WNL.0000000000003771. Epub 2017 Feb 24. PMID 28235817
- [Derived] Delcourt C, Zheng D, Chen X, Hackett M, Arima H, Hata J, Heeley E, Al-Shahi Salman R, Woodward M, Huang Y, Robinson T, Lavados PM, Lindley RI, Stapf C, Davies L, Chalmers J, Anderson CS, Sato S; INTERACT Investigators. Associations with health-related quality of life after intracerebral haemorrhage: pooled analysis of INTERACT studies. J Neurol Neurosurg Psychiatry. 2017 Jan;88(1):70-75. doi: 10.1136/jnnp-2016-314414. Epub 2016 Oct 21. PMID 27919055
- [Derived] Munoz Venturelli P, Wang X, Zahuranec DB, Lavados PM, Stapf C, Lindley R, Delcourt C, Chalmers J, Anderson CS, Robinson TG, Robinson TG; INTERACT2 Investigators. Withdrawal of active treatment after intracerebral haemorrhage in the INTERACT2 study. Age Ageing. 2017 Mar 1;46(2):329-332. doi: 10.1093/ageing/afw187. PMID 27831492
- [Derived] Song L, Sandset EC, Arima H, Heeley E, Delcourt C, Chen G, Yang J, Wu G, Wang X, Lavados PM, Huang Y, Stapf C, Wang J, Robinson TG, Chalmers J, Lindley RI, Anderson CS; INTERACT2 Investigators. Early blood pressure lowering in patients with intracerebral haemorrhage and prior use of antithrombotic agents: pooled analysis of the INTERACT studies. J Neurol Neurosurg Psychiatry. 2016 Dec;87(12):1330-1335. doi: 10.1136/jnnp-2016-313246. Epub 2016 May 13. PMID 27178897
- [Derived] Qiu M, Sato S, Zheng D, Wang X, Carcel C, Hirakawa Y, Sandset EC, Delcourt C, Arima H, Wang J, Chalmers J, Anderson CS; INTERACT Investigators*. Admission Heart Rate Predicts Poor Outcomes in Acute Intracerebral Hemorrhage: The Intensive Blood Pressure Reduction in Acute Cerebral Hemorrhage Trial Studies. Stroke. 2016 Jun;47(6):1479-85. doi: 10.1161/STROKEAHA.115.012382. Epub 2016 May 10. PMID 27165954
- [Derived] Carcel C, Wang X, Sato S, Stapf C, Sandset EC, Delcourt C, Arima H, Robinson T, Lavados P, Chalmers J, Anderson CS; INTERACT2 Investigators*. Degree and Timing of Intensive Blood Pressure Lowering on Hematoma Growth in Intracerebral Hemorrhage: Intensive Blood Pressure Reduction in Acute Cerebral Hemorrhage Trial-2 Results. Stroke. 2016 Jun;47(6):1651-3. doi: 10.1161/STROKEAHA.116.013326. Epub 2016 May 3. PMID 27143274
- [Derived] Delcourt C, Zhang S, Arima H, Sato S, Al-Shahi Salman R, Wang X, Davies L, Stapf C, Robinson T, Lavados PM, Chalmers J, Heeley E, Liu M, Lindley RI, Anderson CS; INTERACT2 investigators. Significance of Hematoma Shape and Density in Intracerebral Hemorrhage: The Intensive Blood Pressure Reduction in Acute Intracerebral Hemorrhage Trial Study. Stroke. 2016 May;47(5):1227-32. doi: 10.1161/STROKEAHA.116.012921. Epub 2016 Apr 12. PMID 27073236
- [Derived] Munoz-Venturelli P, Wang X, Lavados PM, Stapf C, Robinson T, Lindley R, Heeley E, Delcourt C, Chalmers J, Anderson CS; INTERACT2 Investigators. Prophylactic heparin in acute intracerebral hemorrhage: a propensity score-matched analysis of the INTERACT2 study. Int J Stroke. 2016 Jul;11(5):549-56. doi: 10.1177/1747493016641113. Epub 2016 Mar 23. PMID 27009893
- [Derived] Zheng D, Arima H, Sato S, Gasparrini A, Heeley E, Delcourt C, Lo S, Huang Y, Wang J, Stapf C, Robinson T, Lavados P, Chalmers J, Anderson CS; INTERACT2 investigators. Low Ambient Temperature and Intracerebral Hemorrhage: The INTERACT2 Study. PLoS One. 2016 Feb 9;11(2):e0149040. doi: 10.1371/journal.pone.0149040. eCollection 2016. PMID 26859491
- [Derived] Sato S, Delcourt C, Heeley E, Arima H, Zhang S, Al-Shahi Salman R, Stapf C, Woo D, Flaherty ML, Vagal A, Levi C, Davies L, Wang J, Robinson T, Lavados PM, Lindley RI, Chalmers J, Anderson CS; INTERACT2 Investigators. Significance of Cerebral Small-Vessel Disease in Acute Intracerebral Hemorrhage. Stroke. 2016 Mar;47(3):701-7. doi: 10.1161/STROKEAHA.115.012147. Epub 2016 Feb 4. PMID 26846860
- [Derived] Saxena A, Anderson CS, Wang X, Sato S, Arima H, Chan E, Munoz-Venturelli P, Delcourt C, Robinson T, Stapf C, Lavados PM, Wang J, Neal B, Chalmers J, Heeley E; INTERACT2 Investigators. Prognostic Significance of Hyperglycemia in Acute Intracerebral Hemorrhage: The INTERACT2 Study. Stroke. 2016 Mar;47(3):682-8. doi: 10.1161/STROKEAHA.115.011627. Epub 2016 Jan 26. PMID 26814235
- [Derived] Yu S, Arima H, Heeley E, Delcourt C, Krause M, Peng B, Yang J, Wu G, Chen X, Chalmers J, Anderson CS; INTERACT2 Investigators. White blood cell count and clinical outcomes after intracerebral hemorrhage: The INTERACT2 trial. J Neurol Sci. 2016 Feb 15;361:112-6. doi: 10.1016/j.jns.2015.12.033. Epub 2015 Dec 22. PMID 26810526
- [Derived] Moullaali TJ, Sato S, Wang X, Rabinstein AA, Arima H, Carcel C, Chen G, Robinson T, Heeley E, Chan E, Delcourt C, Stapf C, Cordonnier C, Lindley RI, Chalmers J, Anderson CS; INTERACT Investigators. Prognostic significance of delayed intraventricular haemorrhage in the INTERACT studies. J Neurol Neurosurg Psychiatry. 2017 Jan;88(1):19-24. doi: 10.1136/jnnp-2015-311562. Epub 2016 Jan 8. PMID 26746184
- [Derived] Wang X, Arima H, Yang J, Zhang S, Wu G, Woodward M, Munoz-Venturelli P, Lavados PM, Stapf C, Robinson T, Heeley E, Delcourt C, Lindley RI, Parsons M, Chalmers J, Anderson CS; INTERACT2 Investigators. Mannitol and Outcome in Intracerebral Hemorrhage: Propensity Score and Multivariable Intensive Blood Pressure Reduction in Acute Cerebral Hemorrhage Trial 2 Results. Stroke. 2015 Oct;46(10):2762-7. doi: 10.1161/STROKEAHA.115.009357. Epub 2015 Aug 11. PMID 26265125
- [Derived] Sato S, Arima H, Heeley E, Hirakawa Y, Delcourt C, Lindley RI, Robinson T, Huang Y, Morgenstern L, Stapf C, Wang J, Chalmers J, Anderson CS; INTERACT2 Investigators. Off-Hour Admission and Outcomes in Patients with Acute Intracerebral Hemorrhage in the INTERACT2 Trial. Cerebrovasc Dis. 2015;40(3-4):114-20. doi: 10.1159/000434690. Epub 2015 Jul 18. PMID 26202097
- [Derived] Heeley E, Anderson CS, Woodward M, Arima H, Robinson T, Stapf C, Parsons M, Lavados PM, Huang Y, Wang Y, Crozier S, Parry-Jones A, Wang J, Chalmers J; INTERACT2 Investigators. Poor utility of grading scales in acute intracerebral hemorrhage: results from the INTERACT2 trial. Int J Stroke. 2015 Oct;10(7):1101-7. doi: 10.1111/ijs.12518. Epub 2015 Jun 4. PMID 26044442
- [Derived] Wang X, Arima H, Al-Shahi Salman R, Woodward M, Heeley E, Stapf C, Lavados PM, Robinson T, Huang Y, Wang J, Delcourt C, Anderson CS. Rapid Blood Pressure Lowering According to Recovery at Different Time Intervals after Acute Intracerebral Hemorrhage: Pooled Analysis of the INTERACT Studies. Cerebrovasc Dis. 2015;39(3-4):242-8. doi: 10.1159/000381107. Epub 2015 Mar 25. PMID 25823544
- [Derived] Wang X, Arima H, Heeley E, Delcourt C, Huang Y, Wang J, Stapf C, Robinson T, Woodward M, Chalmers J, Anderson CS; INTERACT2 Investigators. Magnitude of blood pressure reduction and clinical outcomes in acute intracerebral hemorrhage: intensive blood pressure reduction in acute cerebral hemorrhage trial study. Hypertension. 2015 May;65(5):1026-32. doi: 10.1161/HYPERTENSIONAHA.114.05044. Epub 2015 Mar 23. PMID 25801872
- [Derived] Yang J, Arima H, Wu G, Heeley E, Delcourt C, Zhou J, Chen G, Wang X, Zhang S, Yu S, Chalmers J, Anderson CS; INTERACT Investigators. Prognostic significance of perihematomal edema in acute intracerebral hemorrhage: pooled analysis from the intensive blood pressure reduction in acute cerebral hemorrhage trial studies. Stroke. 2015 Apr;46(4):1009-13. doi: 10.1161/STROKEAHA.114.007154. Epub 2015 Feb 24. PMID 25712944
- [Derived] Chan E, Anderson CS, Wang X, Arima H, Saxena A, Moullaali TJ, Heeley E, Delcourt C, Wu G, Wang J, Chen G, Lavados PM, Stapf C, Robinson T, Chalmers J, Huang Y; INTERACT2 Investigators. Significance of intraventricular hemorrhage in acute intracerebral hemorrhage: intensive blood pressure reduction in acute cerebral hemorrhage trial results. Stroke. 2015 Mar;46(3):653-8. doi: 10.1161/STROKEAHA.114.008470. Epub 2015 Feb 12. PMID 25677598
- [Derived] Priglinger M, Arima H, Anderson C, Krause M; INTERACT Investigators. No relationship of lipid-lowering agents to hematoma growth: pooled analysis of the intensive blood pressure reduction in acute cerebral hemorrhage trials studies. Stroke. 2015 Mar;46(3):857-9. doi: 10.1161/STROKEAHA.114.007664. Epub 2015 Feb 5. PMID 25657175
- [Derived] Sato S, Heeley E, Arima H, Delcourt C, Hirakawa Y, Pamidimukkala V, Li Z, Tao Q, Xu Y, Hennerici MG, Robinson T, Tzourio C, Lindley RI, Chalmers J, Anderson CS; INTERACT Investigators; Anderson CS, Huang Y, Wang JG, Arima H, Neal B, Peng B, Heeley E, Skulina C, Parsons MW, Kim JS, Tao QL, Li YC, Jiang JD, Tai LW, Zhang LJ, Xu E, Cheng Y, Heritier S, Morgenstern LB, Chalmers J. Higher mortality in patients with right hemispheric intracerebral haemorrhage: INTERACT1 and 2. J Neurol Neurosurg Psychiatry. 2015 Dec;86(12):1319-23. doi: 10.1136/jnnp-2014-309870. Epub 2015 Jan 14. PMID 25589782
- [Derived] Wang X, Arima H, Al-Shahi Salman R, Woodward M, Heeley E, Stapf C, Lavados PM, Robinson T, Huang Y, Wang J, Delcourt C, Anderson CS; INTERACT Investigators. Clinical prediction algorithm (BRAIN) to determine risk of hematoma growth in acute intracerebral hemorrhage. Stroke. 2015 Feb;46(2):376-81. doi: 10.1161/STROKEAHA.114.006910. Epub 2014 Dec 11. PMID 25503550
- [Derived] Radholm K, Arima H, Lindley RI, Wang J, Tzourio C, Robinson T, Heeley E, Anderson CS, Chalmers J; INTERACT2 Investigators. Older age is a strong predictor for poor outcome in intracerebral haemorrhage: the INTERACT2 study. Age Ageing. 2015 May;44(3):422-7. doi: 10.1093/ageing/afu198. Epub 2014 Dec 13. PMID 25497513
- [Derived] Manning L, Hirakawa Y, Arima H, Wang X, Chalmers J, Wang J, Lindley R, Heeley E, Delcourt C, Neal B, Lavados P, Davis SM, Tzourio C, Huang Y, Stapf C, Woodward M, Rothwell PM, Robinson TG, Anderson CS; INTERACT2 investigators. Blood pressure variability and outcome after acute intracerebral haemorrhage: a post-hoc analysis of INTERACT2, a randomised controlled trial. Lancet Neurol. 2014 Apr;13(4):364-73. doi: 10.1016/S1474-4422(14)70018-3. Epub 2014 Feb 13. PMID 24530176
- [Derived] Chen G, Arima H, Wu G, Heeley E, Delcourt C, Zhang P, Rabinstein AA, Robinson T, Stapf C, Huang Y, Song L, Yang J, Wang X, Li Q, Chen X, Chalmers J, Anderson C; INTERACT2 Investigators. Subarachnoid extension of intracerebral hemorrhage and 90-day outcomes in INTERACT2. Stroke. 2014 Jan;45(1):258-60. doi: 10.1161/STROKEAHA.113.003524. Epub 2013 Oct 22. PMID 24149007
- [Derived] Anderson CS, Heeley E, Huang Y, Wang J, Stapf C, Delcourt C, Lindley R, Robinson T, Lavados P, Neal B, Hata J, Arima H, Parsons M, Li Y, Wang J, Heritier S, Li Q, Woodward M, Simes RJ, Davis SM, Chalmers J; INTERACT2 Investigators. Rapid blood-pressure lowering in patients with acute intracerebral hemorrhage. N Engl J Med. 2013 Jun 20;368(25):2355-65. doi: 10.1056/NEJMoa1214609. Epub 2013 May 29. PMID 23713578
- [Derived] Delcourt C, Stapf C, Tzourio C, Heritier S, Anderson C. [The second (main) phase of an open, randomised, multicentre study to investigate the effectiveness of an INTEnsive blood pressure Reduction in Acute Cerebral hemorrhage Trial (INTERACT2): protocol and baseline characteristics of patients included in France]. Rev Neurol (Paris). 2012 Apr;168(4):321-7. doi: 10.1016/j.neurol.2011.08.010. Epub 2011 Nov 29. French. PMID 22129475

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Blood-Pressure Lowering: Intensive Blood pressure (BP) lowering therapy is given via an intravenous drip for 24 hours. The target is to reach a systolic BP <140mmHg within 1 hour.
  Blood pressure management policies : The trial is an assessment of BP lowering management strategies, using routinely available drugs. There is some flexibility in the use of particular BP lowering agents to achieve BP targets.
- Guideline-Recommended Blood-Pressure Lowering: Patients will receive management of BP that is based on a standard guideline, as published by the American Heart Association (AHA). The attending clinician may consider commencing BP treatment if the systolic level is greater than 180 mmHg, however and the first line treatment will be oral (including nasogastric if required) and/or transdermal routes. Should control of systolic BP not be achieved via these routes, intravenous treatment may be started until the target systolic BP of 180 mmHg is achieved.
  Blood pressure management policies : The trial is an assessment of BP lowering management strategies, using routinely available drugs. There is some flexibility in the use of particular BP lowering agents to achieve BP targets.
Period: Overall Study
Arm/Group | Intensive Blood-Pressure Lowering | Guideline-Recommended Blood-Pressure Lowering
Started | 1403 | 1436
Completed | 1394 | 1421
Not Completed | 9 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Blood-Pressure Lowering | Guideline-Recommended Blood-Pressure Lowering | Total
Number analyzed (Participants) | 1403 | 1436 | 2839
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 797 | 770 | 1567
  >=65 years | 606 | 666 | 1272
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (13.1) | 64.1 (12.6) | 63.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 505 | 554 | 1059
  Male | 898 | 882 | 1780
Region of Enrollment [Number; unit: participants]
  Argentina | 2 | 2 | 4
  Australia | 33 | 40 | 73
  Austria | 35 | 28 | 63
  Belgium | 6 | 6 | 12
  Brazil | 8 | 9 | 17
  Chile | 17 | 12 | 29
  China | 950 | 976 | 1926
  Finland | 19 | 17 | 36
  France | 109 | 112 | 221
  Germany | 70 | 71 | 141
  Hong Kong | 0 | 1 | 1
  India | 48 | 49 | 97
  Italy | 19 | 28 | 47
  Netherlands | 1 | 1 | 2
  Norway | 2 | 3 | 5
  Pakistan | 5 | 4 | 9
  Portugal | 12 | 10 | 22
  Spain | 25 | 25 | 50
  Switzerland | 2 | 1 | 3
  United Kingdom | 35 | 35 | 70
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: A Composite of Death or Dependency, With Dependency Being Defined by a Score of 3 to 5 on the Modified Rankin Scale (mRS)
Time Frame: 90 days
Population: In the intensive group 12 patients were alive at 90 days but missing data on mRS (required for primary outcome), and 9 patients in the guideline group
Measure: Number; unit: participants
Arm/Group | Intensive Blood-Pressure Lowering | Guideline-Recommended Blood-Pressure Lowering
Number analyzed (Participants) | 1382 | 1412
participants | 719 | 785

2. Secondary Outcome: Death at 90 Days
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Intensive Blood-Pressure Lowering | Guideline-Recommended Blood-Pressure Lowering
Number analyzed (Participants) | 1394 | 1421
participants | 166 | 170

ADVERSE EVENTS:
Description: Adverse events were not collected, only Serious Adverse Events.
Arm/Group | Intensive Blood-Pressure Lowering | Guideline-Recommended Blood-Pressure Lowering
Serious Adverse Events (participants affected / at risk) | 324/1399 | 329/1430
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Blood-Pressure Lowering (N=1399) | Guideline-Recommended Blood-Pressure Lowering (N=1430)
Direct effects of primary ICH event (General disorders) | 143 | 154
ICH (Vascular disorders) | 5 | 7
Ischaemic/undifferentiated stroke (Vascular disorders) | 9 | 8
Acute MI/coronary event/other (Cardiac disorders) | 5 | 6
Other vascular disease (Vascular disorders) | 15 | 16
Other cardiac disease (Cardiac disorders) | 24 | 27
Renal failure (Renal and urinary disorders) | 6 | 11
Severe hypotension (Vascular disorders) | 8 | 12
Respiratory infections (Infections and infestations) | 66 | 77
Sepsis (includes other infections) (Infections and infestations) | 26 | 24
Non-vasular medical (General disorders) | 52 | 50
Non-vasular injury (including fracture) (Injury, poisoning and procedural complications) | 107 | 96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes